CLINICAL TRIAL: NCT01267162
Title: Long-term Observational Study on Anti-HBV Effect of Tenofovir Disoproxil Fumarate (TDF) and Resistance Surveillance in Asian-American Adult Patients Formerly Participating Gilead 123 Studies
Brief Title: Long-term Study on Anti-HBV Effect of Tenofovir and Resistance Surveillance in Asian-American Adult Patients
Status: Completed | Type: Observational
Sponsor: Medical Procare PLLC (Other)
Responsible Party: Sponsor
Other Study IDs: IN-US-174-0156
Record Dates: First submitted 2010-12-23; First posted 2010-12-28 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2016-03

CONDITIONS: Chronic Hepatitis B
Keywords: CHB
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- TDF Treatment

SUMMARY:
This is a Phase IV, open-label, single-arm, 96 week community-based observational study evaluating the antiviral efficacy, safety, and tolerability of TDF in HBV mono-infected Asian-American adults who had completed 48 week treatment with Tenofovir in Gilead 174-0123 study. The primary objective of this study is to evaluate the long-term antiviral efficacy of tenofovir DF 300 mg once daily in these patients. The secondary objectives are to evaluate the safety and tolerability of TDF including the biochemical and virological responses to TDF, the incidence of drug resistance mutations in these patients The duration of treatment in this study is total of three Years (144 weeks) on TDF.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, Asian-American, who have participated and completed the study, qualify the following criteria, and remain on TDF treatment without severe treatment-related AEs, and with available retrospective lab results as summarized in Appendix 2.
* 18 through 75 years of age, inclusive
* Willing to participate in the present study and able to provide written informed consent
* Continuation of HBV treatment is indicated. That is for HBeAg-positive subjects, HBeAg remain positive or HBeAg becomes negative but still has detectable DNA by the PCR method; and for HBeAg-negative subjects, HBV DNA is either detectable or undetectable by the PCR method
* No clinical or virologic evidence of anti-HBV resistance to TDF treatment at the time of entering tests (i.e., TDF treatment week 48 lab tests by the 123 study)
* Estimated glomerular filtration rate (creatinine clearance) ≥ 60 mL/min/1.73m2 by the

Cockcroft-Gault equation:

(140-age in years) (body weight [kg]) (72) (serum creatinine [mg/dl]) [Note: multiply estimated rate 0. by 85 for women; use actual body weight]

• Adequate hematologic function (absolute neutrophil count ≥ 1,500/mm3; hemoglobin ≥ 10.0 g/dL)

Exclusion Criteria:

* Pregnant women, and women who are breast feeding or who believe they may wish to become pregnant during the course of the study.
* Males and females of reproductive potential who are not willing to use an effective method of contraception during the study. For males, condoms should be used and for females, a barrier contraception method should be used in combination with one other form of contraception.
* Willing and able to provide written informed consent
* Decompensated liver disease defined as direct (conjugated) bilirubin ≥ 1.2 ULN; PT ≥ 1.2 ULN, platelets ≤ 150,000/mm3, or serum albumin ≤ 3.5 g/dL
* Prior history of clinical hepatic decompensation (e.g., ascites, jaundice, encephalopathy) or variceal hemorrhage
* Serum α-fetoprotein ≥ 50 ng/mL
* Evidence of hepatocellular carcinoma (HCC)
* Co-infection with HIV, HCV, or HDV
* History of significant renal disease (e.g., nephrotic syndrome, renal dysgenesis, polycystic kidney disease, congenital nephrosis, acute tubular necrosis, other renal disease)
* History of significant bone disease (e.g., osteomalacia, chronic osteomyelitis, osteogenesis imperfecta, osteochondroses, multiple bone fractures)
* Significant cardiovascular, pulmonary or neurological disease
* Evidence of a gastrointestinal malabsorption syndrome that may interfere with absorption of orally administered medications
* History of solid organ or bone marrow transplantation
* Ongoing therapy with any of the following: Nephrotoxic agents
* Parenteral aminoglycoside antibiotics (e.g., gentamicin, tobramycin, amikacin)
* Cidofovir
* Cisplatin
* Foscarnet
* IV amphotericin B
* IV pentamidine
* Oral or IV ganciclovir
* Cyclosporine
* Tacrolimus
* IV vancomycin
* Chronic daily non-steroidal anti-inflammatory drug therapy
* Competitors of renal excretion (e.g., probenecid) Systemic chemotherapeutic agents
* Systemic corticosteroids
* Interleukin-2 (IL-2) and other immunomodulating agents

Investigational agents (except with the expressed approval of the lead investigators) Administration of any of the above medications must be discontinued at least 30 days prior to the Baseline Visit and for the duration of the study period.

* Known hypersensitivity to the study drugs, the metabolites or formulation excipients
* Any other condition (including alcohol or substance abuse) or prior therapy that, in the opinion of the Investigators, would make the subject unsuitable for the study or unable to comply with dosing requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult infected with chronic hepatitis B
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2010-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
HBV DNA suppression | in three years
safety use of TDF | in three years
  including elevation of creatine or decrease in GFR, TDF resistance

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Asian Pacific Liver Center of St. Vincent Medical Center, Los Angeles, California
  - San Jose Gastroenterology, San Jose, California
  - Dreamworks Endoscopy, Flushing, New York
  - Dr. Calvin Pan's Flushing Office, Flushing, Queens, New York
  - Xiaoli Ma, PC, Philadelphia, Pennsylvania